CLINICAL TRIAL: NCT03631407
Title: A Phase 2 Trial to Evaluate the Safety and Efficacy of Vicriviroc (MK-7690) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Microsatellite Stable (MSS) Colorectal Cancer (CRC)
Brief Title: Safety and Efficacy of Vicriviroc (MK-7690) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Microsatellite Stable (MSS) Colorectal Cancer (CRC) (MK-7690-046)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7690-046; MK-7690-046 (Other: MSD)
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Neoplasms
Keywords: programmed cell death 1 (PD-1, PD1 ); programmed cell death ligand 1 (PD-L1, PDL1); microsatellite stable (MSS) colorectal cancer (CRC); chemokine receptor type 5 (CCR5)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body; Spinocerebellar Degenerations | interventions — vicriviroc; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) (Experimental): Participants receive vicriviroc 150 mg tablets per os (PO) every day (QD) of each 21-day cycle up to 35 cycles and pembrolizumab 200 mg as a 30-minute intravenous (IV) infusion on Day 1 of each 21 day cycle up to 35 cycles (cycle length: 21 days).
  Interventions: Drug: Vicriviroc; Biological: Pembrolizumab
- Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg) (Experimental): Participants receive vicriviroc 250 mg tablets PO QD of each 21-day cycle up to 35 cycles and pembrolizumab 200 mg as a 30-minute IV infusion on Day 1 of each 21 day cycle up to 35 cycles (cycle length: 21 days).
  Interventions: Drug: Vicriviroc; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Vicriviroc — Vicriviroc tablets administered orally, QD at dose level 1 or 2.
  Other Names: MK-7690
Biological: Pembrolizumab — Pembrolizumab administered by IV infusion at 200 mg every 3 weeks (Q3W), given on cycle day 1.
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
This trial will evaluate the safety and efficacy of vicriviroc (MK-7690) at 2 dose levels in combination with pembrolizumab (MK-3475) in participants with advanced/metastatic microsatellite stable (MSS) colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically proven locally advanced unresectable or metastatic CRC.
* Have locally confirmed MSS CRC.
* Have been previously treated with standard therapies, which must include fluoropyrimidine, oxaliplatin, and irinotecan, and have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit.
* Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days of starting study intervention.
* Male participants must agree to use contraception and refrain from donating sperm for at least 120 days after the last dose of study intervention.
* Female participants must be not pregnant and not breastfeeding. Further, a female participant must either not be a woman of childbearing potential (WOCBP) or, if a WOCBP, agree to use contraception during the treatment period and for at least 120 days after the last dose of study intervention.
* Have adequate organ function.

Exclusion Criteria:

* Have a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Have severe hypersensitivity reaction to treatment with any monoclonal antibody or components of the study interventions.
* Have an active autoimmune disease requiring systemic treatment in the past 2 years, except vitiligo or resolved childhood asthma/atopy.
* Have a history of vasculitis.
* Have an active infection requiring systemic therapy.
* Have symptomatic ascites or pleural effusion.
* Have interstitial lung disease requiring oral or IV glucocorticoids.
* Have a history of pneumonitis (noninfectious) that required steroids, or has current pneumonitis.
* Have a known history of human immunodeficiency virus (HIV) infection.
* Have a known history of hepatitis B or known active hepatitis C virus infection.
* Have a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, make administration of the study interventions hazardous, or make it difficult to monitor adverse events.
* Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with study requirements.
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study intervention.
* Are a WOCBP who has a positive urine pregnancy test within 72 hours before randomization or treatment allocation.
* Have undergone major surgery and have not recovered adequately from any toxicity and/or complications from the intervention before starting study intervention.
* Have a seizure disorder requiring ongoing antiseizure therapy or with any condition that, in the judgment of the investigator, is likely to increase the risk of seizure (e.g., CNS malignancy or toxoplasmosis).
* Have known gastrointestinal (GI) disease such as esophageal, gastric, or duodenal ulceration or inflammatory bowel disease, or history of GI surgery.
* Are using any drug (therapeutic or recreational), or withdrawal thereof, that poses an increased risk of convulsions.
* Have had an allogeneic tissue/solid organ transplant.
* Have received prior therapy with vicriviroc or other CCR5 antagonist (e.g., maraviroc) or have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent.
* Have been treated with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137).
* Have received prior systemic anticancer therapy, including investigational agents, or has used an investigational device within 28 days before the first dose of study intervention.
* Have received prior radiotherapy (not to target lesions) within 2 weeks of start of study intervention.
* Are expected to require any other form of antineoplastic therapy while on study.
* Have a diagnosis of immunodeficiency, is receiving chronic systemic steroid therapy in excess of replacement doses (prednisone ≤10 mg/day is acceptable), or is taking any other form of immunosuppressive medication within 7 days before the first dose of the study intervention.
* Have received a live-virus vaccine within 30 days before the first dose of the study intervention.
* Are currently participating in or have participated in a study of an investigational agent, or have used an investigational device within 28 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- United States (6):
  - Honor Health ( Site 0103), Scottsdale, Arizona
  - California Cancer Associates for Research & Excellence ( Site 0100), Encinitas, California
  - California Cancer Associates for Research & Excellence ( Site 0102), Fresno, California
  - Florida Cancer Specialists (South Region) - Research Office ( Site 7001), Fort Myers, Florida
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute ( Site 7000), Nashville, Tennessee
  - Baylor Scott & White Medical Center - Temple ( Site 0104), Temple, Texas
- Canada (2):
  - Cross Cancer Institute ( Site 0201), Edmonton, Alberta
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0204), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bessudo A, Haseeb AM, Reeves JA, Zhu X, Wong L, Giranda V, Suttner L, Liu F, Chatterjee M, Sharma S. Safety and Efficacy of Vicriviroc (MK-7690) in Combination With Pembrolizumab in Patients With Advanced or Metastatic Microsatellite Stable Colorectal Cancer. Clin Colorectal Cancer. 2024 Sep;23(3):285-294. doi: 10.1016/j.clcc.2024.05.003. Epub 2024 May 13. PMID 38942693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 participants with advanced/metastatic microsatellite stable (MSS) colorectal cancer (CRC) were randomized to receive vicriviroc in combination with pembrolizumab in this study. Qualified participants were randomized 1:1 to receive vicriviroc (150 mg or 250 mg) in combination with pembrolizumab (200 mg Q3W) using an interactive response technology (IRT).
Groups:
- Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg): Participants received vicriviroc 150 mg tablets per os (PO) every day (QD) of each 21-day cycle up to 35 cycles and pembrolizumab 200 mg administered as a 30-minute intravenous (IV) infusion on Day 1 of each 21 day cycle up to 35 cycles (cycle length: 21 days).
- Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg): Participants received vicriviroc 250 mg tablets per os (PO) every day (QD) of each 21-day cycle up to 35 cycles and pembrolizumab 200 mg administered as a 30-minute intravenous (IV) infusion on Day 1 of each 21 day cycle up to 35 cycles (cycle length: 21 days).
Period: Overall Study
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Started | 21 | 20
Treated | 20 | 20
Completed | 1 | 0
Not Completed | 20 | 20
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Sponsor Decision | 0 | 2
Not completed — Death | 16 | 16
Not completed — Randomized by mistake without study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg) | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (12.1) | 60.4 (11.4) | 59.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 17 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)
Description: Objective response rate (ORR) was defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by the investigator. ORR was estimated and analyzed using Clopper-Pearson interval.
Time Frame: Up to ~32 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, and had a baseline scan with measurable disease per investigator's assessment per RECIST 1.1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9]

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLTs were assessed during the first cycle (21 days) & were defined as: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia, Gr 4 thrombocytopenia of any duration, Gr 3 thrombocytopenia associated with bleeding; nonhematologic adverse event (AE) ≥ Gr 3 (with exceptions); Gr 3 or 4 nonhematologic lab abnormality (if medical intervention was required, lead to hospitalization, or persisted for >72 hours); Gr 3 or 4 febrile neutropenia; inability to receive ≥75% of the planned vicriviroc dose because of drug-related tolerability; drug-related toxicity that caused a >2 week delay in Cycle 2 initiation; elevated aspartate aminotransferase or alanine aminotransferase lab value that is >3× upper limit of normal (ULN) & an elevated total bilirubin value >2× ULN & an alkaline phosphatase value <2× ULN, in which no alternative reasons were found.
Time Frame: Up to Day 21 of Cycle 1 (each cycle is 21 days)
Population: The analysis population consisted of all treated participants who received at least one dose of study drug and finished Cycle 1 without a DLT or experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 18 | 18
Participants | 0 | 2

3. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one AE was assessed.
Time Frame: Up to ~28 months
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed
Time Frame: Up to ~25 months
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Participants | 4 | 7

5. Secondary Outcome: Objective Response Rate (ORR) Based on Modified Response Evaluation Criteria in Solid Tumors 1.1 for Immune-based Therapeutics (iRECIST)
Description: An objective response rate was defined as the percentage of participants who experienced an immune-based complete response (iCR: disappearance of all target lesions) or immune-based partial response (iPR: at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experienced an iCR or iPR using immune-based therapeutics Response Evaluation Criteria in Solid Tumors (iRECIST) per investigator was presented. ORR was estimated and analyzed using Clopper-Pearson interval.
Time Frame: Up to ~32 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, and had a baseline scan with measurable disease per investigator's assessment per modified iRECIST.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Percentage of Participants | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9]

6. Secondary Outcome: Progression-Free Survival (PFS) Based on Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from the first dose of study treatment to the date of the first documentation of disease progression, as determined by investigator per RECIST 1.1 or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: Up to ~32 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Months | 2.1 [1.8 to 3.0] | 2.1 [1.6 to 3.9]

7. Secondary Outcome: PFS Based on Modified Response Evaluation Criteria in Solid Tumors 1.1 for Immune-based Therapeutics (iRECIST)
Description: PFS was defined as the time from the first dose of study treatment to the date of the first documentation of disease progression, as determined by investigator per modified iRECIST or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: Up to ~32 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Months | 4.0 [2.7 to 5.6] | 4.9 [3.1 to 8.0]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of study treatment until death from any cause.
Time Frame: Up to ~32 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, and had a baseline scan with measurable disease per investigator's assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
Months | 4.6 [2.7 to 12.6] | 5.3 [3.2 to 8.0]

9. Secondary Outcome: Plasma Area Under the Concentration Time-Curve From 0 to 8 Hours (AUC 0-8hrs) of Vicriviroc
Description: Plasma vicriviroc concentration was quantified for each arm to determine AUC 0-8hrs, defined as the area under the concentration vs. time curve for vicriviroc from 0 to 8 hours.
Time Frame: Pre-dose, 1, 2, 4, and 8 hours after vicriviroc administration on Cycle 1 (each cycle= 21-days) Day 1, Cycle 2 Day 1.
Population: The analysis population consisted of all participants who received at least 1 treatment and who contributed blood samples for analysis of AUC 0-8hrs. Per protocol, AUC 0-8hrs was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
hr*ng/mL
  Cycle 1: number analyzed (Participants) | 19 | 19
  Cycle 1 | 2600 (30.6) | 4790 (62.6)
  Cycle 2: number analyzed (Participants) | 16 | 13
  Cycle 2 | 4940 (46.4) | 10600 (84.4)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Vicriviroc
Description: Plasma vicriviroc concentration was quantified for each arm to determine Cmax, defined as the maximum observed concentration of vicriviroc in plasma.
Time Frame: Pre-dose, 1, 2, 4, and 8 hours after vicriviroc administration on Cycle 1 (each cycle= 21-days) Day 1, Cycle 2 Day 1.
Population: The analysis population consisted of all participants who received at least 1 treatment and who contributed blood samples for analysis of Cmax. Per protocol, Cmax was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 20 | 20
ng/mL
  Cycle 1 | 656 (37.1) | 1130 (65.3)
  Cycle 2: number analyzed (Participants) | 17 | 14
  Cycle 2 | 955 (45.6) | 1940 (72.7)

11. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Vicriviroc
Description: Plasma vicriviroc concentration was quantified for each arm to determine Ctrough, defined as the minimum plasma concentration of vicriviroc observed after administration and just before the subsequent dose.
Time Frame: Pre-dose, and 1, 2, 4, and 8 hours after vicriviroc administration on Cycle 1 (each cycle= 21-days) Day 1; Cycle 3 Day 21.
Population: The analysis population consisted of all participants who received at least 1 treatment and who contributed blood samples for analysis of Ctrough. Per protocol, Ctrough was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
Number analyzed (Participants) | 15 | 11
ng/mL
  Cycle 1 | 338 (102.3) | 468 (162.6)
  Cycle 3: number analyzed (Participants) | 8 | 7
  Cycle 3 | 217 (61.9) | 635 (62.4)

ADVERSE EVENTS:
Time Frame: For AEs: Up to ~28 months. All-cause mortality (ACM): Up to ~32 months.
Description: All-cause mortality includes all randomized participants. Safety includes participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg)
All-Cause Mortality (participants affected / at risk) | 19/21 | 17/20
Serious Adverse Events (participants affected / at risk) | 12/20 | 10/20
Other Adverse Events (participants affected / at risk) | 14/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) (N=20) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg) (N=20)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Visual field defect (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2)
Death (General disorders) | 1 (1) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vicriviroc QD at Dose Level 1 (150 mg) + Pembrolizumab (200 mg) (N=20) | Vicriviroc QD at Dose Level 2 (250 mg) + Pembrolizumab (200 mg) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (8)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (6)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (6) | 4 (4)
Chills (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (7) | 8 (8)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (6) | 6 (8)
Alanine aminotransferase increased (Investigations) | 3 (3) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 4 (4) | 3 (4)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 6 (7)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03631407/Prot_SAP_000.pdf